CLINICAL TRIAL: NCT04123418
Title: A Phase I, Open-label, Multicenter, Study of WVT078 in Subjects With Relapsed and/or Refractory Multiple Myeloma
Brief Title: A Study of WVT078 in Patients With Multiple Myeloma (MM)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision was made for business reasons and was not based on any safety or tolerability concerns
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CWVT078A12101
Record Dates: First submitted 2019-10-02; First posted 2019-10-10 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma (MM)
Keywords: Multiple Myeloma, phase 1
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- WVT078 in Multiple Myeloma (MM) patients (Experimental): Dose escalation study to determine Maximum Tolerated Dose (MTD)/ Recommended Dose (RD) in adult patients with relapsed and/or refractory Multiple Myeloma (MM)
  Interventions: Biological: WVT078
- WVT078 in combination with WHG626 in Multiple Myeloma (MM) patients (Experimental): Dose escalation study to determine Maximum Tolerated Dose (MTD)/ Recommended Dose (RD) in adult patients with relapsed and/or refractory Multiple Myeloma (MM)
  Interventions: Biological: WVT078; Drug: WHG626

INTERVENTIONS:
Biological: WVT078 — WVT078 will be administered IV (intravenously) in a dose escalation schedule
Drug: WHG626 — WHG626 will be administered orally in a dose escalation schedule
  Arms: WVT078 in combination with WHG626 in Multiple Myeloma (MM) patients

SUMMARY:
The design of a phase I, open-label, dose finding study was chosen in order to establish a safe and tolerated dose of single agent WVT078 alone and in combination with WHG626 in patients relapses and/or refractory Multiple Myeloma (MM)

DETAILED DESCRIPTION:
This first-in-human trial with WVT078 is a dose escalation study whose primary purpose is to characterize the safety, tolerability, and determine recommended dose regimen(s) of WVT078 alone and in combination with WHG626 in subjects with MM who have received two or more standard of care lines of therapy including an IMID, a proteasome inhibitor, and an anti-CD38 agent (if available) and are relapsed and/or refractory to or intolerant of each regimen. In addition, this study will assess preliminary anti-MM response of and characterize the pharmacokinetics and immunogenicity of WVT078 alone and in combination with WHG626. The results of this study will inform the future development of WVT078 alone and in combination with WHG626 as a treatment for relapsed and/or refractory MM.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are relapsed and/or refractory to two or more regimens including an IMID, proteasome inhibitor, and an anti-CD38 agent (if available)

Exclusion Criteria:

* Use of systemic chronic steroid therapy (>or= 10mg/day prednisone or equivalent) or any immunosuppressive therapy within 7 days of first dose of study treatment
* Malignant disease other than being treated on this study
* Active known or suspected autoimmune disease
* Impaired cardiac function or clinically significant cardiac disease
* Treatment with cytotoxic or small molecule antineoplastics or any experimental therapy within 14 days or 5 half-lives whichever is shorter
* Active central nervous system involvement by malignancy or presence of symptomatic CNS metasteses

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLTs) in Cycle 1 | 28 days (first cycle)
  To characterize the safety, tolerability, and determine the recommended dose regimen(s) of WVT078 alone and in combination with WHG626 in subjects with relapsed and/or refractory MM
Frequency of dose interruptions | Up to 28 months
  To characterize the safety, tolerability, and determine the recommended dose regimen(s) of WVT078 alone and in combination with WHG626 in subjects with relapsed and/or refractory MM
Frequency of discontinuations | up to 28 months
  To characterize the safety, tolerability, and determine the recommended dose regimen(s) of WVT078 alone and in combination with WHG626 in subjects with relapsed and/or refractory MM
Frequency of dose reductions | up to 28 months
  To characterize the safety, tolerability, and determine the recommended dose regimen(s) of WVT078 alone and in combination with WHG626 in subjects with relapsed and/or refractory MM
Incidence and severity of AEs and SAEs, including changes in laboratory values, vital signs, ECGs, and CRS/immune-mediated reactions | Up to 31 months
  To characterize the safety, tolerability, and determine the recommended dose regimen(s) of WVT078 alone and in combination with WHG626 in subjects with relapsed and/or refractory MM

SECONDARY OUTCOMES:
Best Overall Response (BOR) | Up to 36 months
  Response assessment per International Myeloma Working Group (IMWG) criteria
Duration of Response (DOR) | Up to 36 months
  Response assessment per International Myeloma Working Group (IMWG) criteria
Progresson Free Survival (PFS) | Up to 36 months
  Response assessment per International Myeloma Working Group (IMWG) criteria
AUC of WVT078 derived from serum concentrations | Up to 28 months
Cmax of WVT078 derived from serum concentrations | Up to 28 months
Cmin of WVT078 derived from serum concentrations | Up to 28 months
Tmax of WVT078 derived from serum concentrations | Up to 28 months
T1/2 of WVT078 derived from serum concentrations | Up to 28 months
Concentration of WVT078 Anti Drug Antibodies (ADA) as measured in serum | Up to 28 months
AUC of WHG626 derived from plasma concentrations | Up to 28 months
Cmax of WHG626 derived from plasma concentrations | Up to 28 months
Cmin of WHG626 derived from plasma concentrations | Up to 28 months
Tmax of WHG626 derived from plasma concentrations | Up to 28 months
T1/2 of WHG626 derived from plasma concentrations | Up to 28 months
AUC of GWQ573 (the active metabolite of WHG626) derived from plasma concentrations | Up to 28 months
Cmax of GWQ573 (the active metabolite of WHG626) derived from plasma concentrations | Up to 28 months
Cmin of GWQ573 (the active metabolite of WHG626) devived from plasma concentrations | Up to 28 months
Tmax of GWQ573 (the active metabolite of WHG626) derived from plasma concentrations | Up to 28 months
T1/2 of GWQ573 (the active metabolite of WHG626) derived from plasma concentrations | Up to 28 months

CONTACTS AND LOCATIONS:
Locations (12):
- United States (3):
  - Emory University School of Medicine-Winship Cancer Institute, Atlanta, Georgia
  - University Of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Novartis Investigative Site, Melbourne, Victoria, Australia
- Germany (2):
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Heidelberg
- Novartis Investigative Site, Tel Aviv, Israel
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Bunkyo Ku, Tokyo, Japan
- Novartis Investigative Site, Oslo, Norway
- Spain (2):
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raab MS, Cohen YC, Schjesvold F, Aardalen K, Oka A, Spencer A, Wermke M, Souza AD, Kaufman JL, Cafro AM, Ocio EM, Doki N, Henson K, Trabucco G, Carrion A, Bender FC, Juif PE, Fessehatsion A, Fan L, Stonehouse JP, Blankenship JW, Granda B, De Vita S, Lu H. Preclinical discovery and initial clinical data of WVT078, a BCMA x CD3 bispecific antibody. Leukemia. 2023 Jun;37(6):1349-1360. doi: 10.1038/s41375-023-01883-3. Epub 2023 Apr 6. PMID 37024520
- See also: CWVT078A12101 Clinical Trial Results Form — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18365
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=3005